CLINICAL TRIAL: NCT04271163
Title: A Phase I Study to Evaluate the Safety and Efficacy of Transcranial Electromagnetic Treatment (TEMT) for the Treatment of Alzheimer's Disease: Extension Study II
Brief Title: Transcranial Electromagnetic Treatment (TEMT) Against Alzheimer's Disease
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: NeuroEM Therapeutics, Inc. (Industry)
Collaborators: Axiom Clinical Research of Florida (Unknown); MegaNano Biotech (Unknown); Invicro, Boston (Unknown); Left Coast Engineering (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EM1000-2
Record Dates: First submitted 2020-02-11; First posted 2020-02-17 (Actual); Last update posted 2020-02-17 (Actual); Status verified 2020-02

CONDITIONS: Alzheimer's Disease
Keywords: Alzheimer's, electromagnetic, cognition, A-beta, tau
MeSH Terms: conditions — Alzheimer Disease; Pick Disease of the Brain

STUDY DESIGN:
Intervention Model Description: Open-Label Pilot Study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: MemorEM — The MemorEM device is self-contained and has been designed for in-home daily electromagnetic treatment in the radiofrequency range to the entire forebrain, allowing for complete mobility and comfort in performing daily activities during treatment. The device has a custom control panel that is powered by a rechargeable battery. This control panel/battery box is worn on the upper arm and wired to specialized emitters in the head cap worn by the subject. Everyday for the 12M treatment period, the subject's caregiver will administer one or two 1-hour treatments (two daily treatments during the first 2M period).

SUMMARY:
This is a second extension of EM 1000-1 wherein mild/moderate AD subjects who participated in the original study have completed participation in a first extension of 4-months. Most of the eight subjects in the original EM 1000-1 and first extension agreed to participate in this second extension study. The time between completion of the first extension and the second extension is 4 months. This second extension study;'s primary objective is to determine the long-term safety and efficacy of 12 months of daily treatment on performance of these AD subjects in the same comprehensive array of cognitive tasks as they performed in the initial 2-month study and 4-month first extension.Secondary objectives include analysis of blood for AD markers and evaluation of safety throughout the treatment period. Upon completion of this 12-month extension, the period between initial treatment and final treatment will be 2-3 years.

DETAILED DESCRIPTION:
The present study is an Open-Label within-patient (single arm) second extension study of the Open-Label 2-month initial study (EM1000-1) and 4M first extension study, wherein most of the original eight AD subjects agree to participate. This present second extension study is intended to continue evaluation of the safety and efficacy of daily Transcranial Electromagnetic Treatment (TEMT) in patients with mild-to-moderate AD for an additional 12 month period, such that the interval between the initial day of treatment and final day of treatment will be 2-3 years.There will be a total of six clinical visits: pre-baseline, baseline, 2-, 5-, 8-, and 12-months. This second extension study will utilize the same MemorEM devices (designated as NSR and not Food and Drug Administration-regulated) as in the first extension studies, but will involve twice daily treatment for the first two months, followed by once-daily treatment thereafter.

Expected Results: The investigators expect that the additional 12 months of daily TEMT will not present any significant side effects or safety issues, as was the case for the initial study and first extension study. The investigators further expect that cognitive measures will be stable and/or improve by the end of the 12M treatment period. In addition, changes in blood/cerebrospinal fluid levels of various beta-amyloid and tau species are anticipated to reflect the primary mechanism of TEMT action -- disaggregation of both A-beta and tau oligomers.

ELIGIBILITY:
Inclusion Criteria:

* Male or female age 63+ years
* Patients diagnosed with mild or moderate stage of Alzheimer's Disease at the beginning of the original treatment study, according to the National Institute of Neurological and Communicative Disorders and Stroke-Alzheimer's Disease and Related Disorders Association (NINCDS-ADRDA) criteria.
* MMSE score 16 to 26 : By the end of Extension Study I, all subjects except for one had MMSE scores above 16.
* Physical clearance for study participation as evaluated by the clinician.
* Caregiver (spouse, family member, etc.) who agrees to and is capable of taking care and being responsible for the participation of the patient in the study (keeping a diary of health measures they collect on the patient at home, logging the patient's condition daily, and assuming responsibility for administering daily in-home treatment). Caregiver to have non-impaired mental abilities and normal motor skills, as determined by the investigators at screening. The definition of caregivers for this study is adults providing unpaid care to relatives or friends to help them take care of themselves in such activities as managing finances, shopping, preparing meals, and going to doctor appointments.
* Agreement to participate in approximately 54 weeks during the study.
* Normal to near-normal vision and hearing with correction as needed (e.g. corrective lenses, hearing aid).
* Fluent in English
* Minimum of 8th grade education
* Head circumference between 53 - 60 cm (to minimize variability in head antenna locations)
* If medicated for AD, then use of cholinesterase inhibitors and/or memantine for at least 3 months, on stable dose for at least 60 days prior to screening, and maintenance on that dose for the period of this study.
* All other non-AD medications must be stable for a period of 4 weeks prior to screening

Exclusion Criteria:

* Severe agitation
* Mental retardation
* Unstable medical condition
* Use of benzodiazepines or barbiturates 2 weeks prior to screening
* Pharmacological immunosuppression
* Participation in a clinical trial with any investigational agent within 6 months prior to study enrollment and no history of immunotherapy research participation
* History of Epileptic Seizures or Epilepsy
* Patients with major depression (not controlled with medication), bipolar disorder or psychotic disorders or any other neurological or psychiatric condition (whether now or in the past). The investigator will obtain this information from available patient medical records, history provided by the patient and caregiver, interview, and neurological exam.
* Alcoholism or drug addiction as defined by (Diagnostic and Statistic Manual of Mental Disorders (DSM)-IV within last 5 years (addicted more than one year and or in remission less than 3 years) or severe sleep deprivation
* Patients with metal implants in the head, (i.e. cochlear implants, implanted brain stimulators, aneurysm clips) with the exception of metal implants in mouth
* Patients with vitamin B12 deficiency, abnormal thyroid function, or personal history of either any clinically defined medical disorder or any clinically defined neurological/psychiatric disorder (other than AD), including (but not limited to):, stroke, brain lesions, , cerebrovascular condition, other neurodegenerative disease, significant head trauma (loss of consciousness greater than half an hour, or related anterograde amnesia), multiple sclerosis; or personal history of previous neurosurgery or brain radiation
* Patients with any signs or symptoms of increased intracranial pressure, as determined in a neurological exam.
* Patients with demonstrated brain micro-hemorrhages (more than 5) at screening
* Patients with a score of 4 or higher on the Hachinski Test
* Patients with a score of 2 or less on the Global Deterioration Scale
* Patients with hypertension that is unresponsive to anti-hypertensive medications
* Patients with a history of migraine headaches occurring more than once a month
* Patients with a history of cancer within last 3 years (basal cell and squamous cell carcinomas will be considered on a case by case basis by investigator)
* Patients chronically taking anticoagulants or anti-platelets (at discretion of PI)
* Pregnant women and women who have the ability to become pregnant
* Patients with compressed hair thickness of more than 5mm (which could increase distance between head antennas and the scalp).
* Cardiac pacemakers
* Implanted medication pumps
* Intracardiac lines
* Significant heart disease

Min Age: 63 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2020-02-10 (Actual); Primary Completion 2021-02-28 (Estimated); Study Completion 2021-03-31 (Estimated)

PRIMARY OUTCOMES:
Alzheimer's Disease Assessment Scale (ADAS)-cog13 score | Changes from baseline ADAS-cog at two, five, eight, and 12 months into treatment
  ADAS-cog is the standard/benchmark test of cognitive performance evaluated in Alzheimer's treatment-based clinical trials. Upper limit is 85 (poor performance) and lower limit is zero (best performance)

SECONDARY OUTCOMES:
Blood (plasma) levels of beta-amyloid1-40 and 1-42, total tau (t-tau), and phospho-tau (p-tau) | Changes from baseline at two, five, eight, and 12 months into treatment
  Blood will be analyzed for beta-amyloid and tau species via specific monoclonal antibody kits
Adverse Event Assessment (Adverse Event Assessment) | Change from baseline Adverse Event Assessment at two, five, eight, and 12 months into treatment.
  AEA will be the primary safety outcome measure
Rey AVLT (Auditory Verbal Learning) score | Changes from baseline Rey AVLT score at two, five, eight, and 12 months into treatment
  This is a secondary cognitive outcome to assess effects of treatment on cognition
Digit span score | Changes from baseline Digit span score at two, five, eight, and 12 months into treatment
  This is a secondary cognitive outcome to assess effects of treatment on cognition
(Mini Mental State Examination (MMSE) score | Changes from baseline MMSE score at two, five, eight, and 12 months into treatment
  This is a secondary cognitive outcome to assess effects of treatment on cognition; maximum (best) score is 30 and minimum (worse) score is zero
Global Deterioration score (GDS) | Changes from baseline GDS score at two, five, eight, and 12 months into treatment
  This is a secondary cognitive outcome to assess effects of treatment on cognition
Trails A & B score | Changes from baseline in Trails A & B scores at two, five, eight, and 12 months into treatment
  This is a secondary cognitive outcome to assess effects of treatment on cognition
Clock draw score | Changes from baseline in clock draw score at two, five, eight, and 12 months into treatment
  This is a secondary cognitive outcome to assess effects of treatment on cognition
MRI Scan (acquisition only) | Change from baseline at 12 months into treatment
  This is a safety outcome to assess any brain consequences of treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Axiom Clinical Research of Florida, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: No
It is not anticipated that Individual Participant Data (IPD) will be shared with other researchers